CLINICAL TRIAL: NCT06733285
Title: Clinical Study to Investigate the Ability of a Stannous Fluoride Toothpaste to Protect From Dentine Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300212
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Toothpaste (Experimental): Participants will dose the toothbrush with a ribbon of test toothpaste, across the full brush head and brush the entire dentition thoroughly for at least 1-timed minute, twice daily (morning and evening) for 2 weeks, making sure to brush the sensitive areas of the two 'test teeth' carefully first.
  Interventions: Drug: Sensodyne Rapid Relief
- Regular Fluoride Toothpaste (Negative Control) (Active Comparator): Participants will dose the toothbrush with a ribbon of regular fluoride toothpaste, across the full brush head and brush the entire dentition thoroughly for at least 1-timed minute, twice daily (morning and evening) for 2 weeks.
  Interventions: Drug: Colgate Cavity Protection

INTERVENTIONS:
Drug: Sensodyne Rapid Relief — Toothpaste containing 0.454 % weight/weight (w/w) SnF2 (1100 parts per million [ppm] fluoride).
  Arms: Test Toothpaste
Drug: Colgate Cavity Protection — A regular fluoride toothpaste containing 1000 ppm fluoride.
  Arms: Regular Fluoride Toothpaste (Negative Control)

SUMMARY:
The purpose of this study is to investigate and characterize the Dentine Hypersensitivity (DH) protection profiles of a 0.454 percent (%) Stannous Fluoride (SnF2) toothpaste and a regular fluoride toothpaste, in response to evaporative air (Schiff sensitivity score) and tactile (tactile threshold in grams [g]) stimuli, with twice daily brushing over 2 weeks.

DETAILED DESCRIPTION:
This will be a single center, randomized, controlled, examiner-blind, 2-arm, stratified, parallel design clinical study in healthy male and female participants, aged 18-70 years, with self-reported and clinically confirmed DH. Participants who meet the required study criteria at screening and baseline will be randomized to one of two study toothpastes: 0.454% SnF2 toothpaste (Test) or a regular fluoride toothpaste (Negative Control). Sufficient participants will be screened to ensure approximately 80 participants are randomized to study toothpaste (approximately 40 participants per group) and approximately 70 participants complete the study (approximately 35 participants per group).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent document confirming the participant has been informed of all pertinent aspects of the study and has given their written consent for study participation before any study procedures are performed.
* Participant is biologically male or female.
* Participant is 18 to 70 years of age, inclusive, at the time of signing the consent form.
* Participant is willing and able to comply with the study visit schedule, toothpaste usage instructions, lifestyle restrictions and other study procedures.
* Participant is in good general, oral and mental health with, in the opinion of the investigator or medically qualified designee, with no clinically significant or relevant abnormalities in self-reported medical history, or upon oral examination that would impact their safety or wellbeing, or the outcomes of the study, if they were to participate in the study, or affect their ability to understand and follow study requirements.

Screening (Visit 1)

* Participants must have:

  1. History of tooth sensitivity lasting more than six months but not more than 10 years (self-reported).
  2. Good general oral health, with a minimum of 20 natural teeth.
  3. Minimum of 2 non-adjacent, accessible teeth (incisors, canines, premolars), in different quadrants, which meet all the following criteria:

     1. Exposed dentine due to facial/cervical erosion or abrasion (that is, tooth wear) or gingival recession (EAR).
     2. Modified Gingival Index (MGI)= 0 directly adjacent to the exposed dentine (that is, the test area only).
     3. Clinical mobility= 0.
     4. Clinically confirmed DH to both tactile and evaporative (air) stimuli: Tactile threshold less than or equal to (<=) 20g and Schiff sensitivity score more than or equal to (>=) 2.

Baseline (Visit 2)

* Participant must have a minimum of two non-adjacent, accessible teeth (incisors, canines, premolars), in different quadrants, with clinically confirmed DH to both tactile and evaporative (air) stimuli at both Screening (Visit 1) and Baseline (Visit 2).

  1. Tactile threshold <= 20g at Screening and Baseline.
  2. Schiff sensitivity score >= 2 at Screening and Baseline.
* The clinical examiner will select two 'test teeth' from those which meet the tactile threshold and Schiff sensitivity score inclusion criteria at both Screening and Baseline.

Exclusion Criteria:

* Participant is an employee of the investigator site directly involved in the conduct of the study, or an employee of the investigator site otherwise supervised by the investigator, or a member of their immediate family.
* Participant is an employee of the sponsor directly involved in the conduct of the study or a member of their immediate family.
* Female participant who is pregnant or intending to become pregnant during the study (self-reported).
* Female participant who is breastfeeding (self-reported).
* Participant with known or suspected intolerance or hypersensitivity to the study products, any of their stated ingredients or closely related compounds (self-reported).
* Participant with a recent history (within the last year) of alcohol or other substance abuse (self-reported).
* Participant is participating in or has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days of Screening (Visit 1) or plans to participate in other studies (including non-medicinal studies) during this study.
* Participant has participated in a tooth sensitivity study within 8 weeks of Screening (Visit 1).
* Participant is currently using an oral care product indicated for DH relief or care of sensitive teeth or has used such a product within 8 weeks of Screening (Visit 1).
* Participant takes daily doses of medications/treatments which, in the opinion of the investigator or medically qualified designee, could interfere with their perception of tooth sensitivity (for example, analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilizers, antidepressants, mood-altering and anti-inflammatory drugs).
* Screening (Visit 1): Participant has taken antibiotics in the 2 weeks prior to Screening (Visit 1).
* Baseline (Visit 2): Participant has taken antibiotics in the 2 weeks prior to Baseline (Visit 2), that is, during the acclimatization period.
* Participant takes daily doses of a medication which, in the opinion of the investigator or medically qualified designee, is causing xerostomia.
* Participant requires antibiotic prophylaxis for dental procedures.
* Participant has had professional tooth de-sensitizing treatment within 8 weeks of Screening (Visit 1).
* Participant has had a tooth bleaching procedure within 8 weeks of Screening (Visit 1).
* Participant has had dental prophylaxis within 4 weeks of Screening (Visit 1).
* Participant has had treatment for periodontal disease (including surgery) within 12 months of Screening (Visit 1).
* Participant has had scaling or root planning within 3 months of Screening (Visit 1).
* Participant with gross periodontal disease.
* Participant with a tongue or lip piercing.
* Participant with evidence of gross intra-oral neglect or the need for extensive dental therapy.
* Participant with a fixed or removable partial prosthesis which, in the opinion of the investigator or dentally qualified designee, could impact study outcomes.
* Participant with multiple dental implants which, in the opinion of the investigator or dentally qualified designee, could impact study outcomes.
* Participant has had orthodontic treatment (fixed or removable orthodontic braces/bands) within 6 months of Screening (Visit 1).
* Participant with a fixed or removable orthodontic retainer which, in the opinion of the investigator or dentally qualified designee, could impact study outcomes (for example, participant who is an intermittent user of a removable orthodontic retainer). Note: Teeth involved in a fixed orthodontic retainer may be used as 'test teeth' if, in the opinion of the investigator or dentally qualified designee, their selection would not impact study outcomes.
* Specific Dentition Exclusions for 'Test teeth':

  1. Tooth with evidence of current/recent dental caries.
  2. Tooth having had (self-reported) treatment for dental caries within 12 months of Screening (Visit 1).
  3. Tooth with exposed dentine and deep, defective, or facial restorations.
  4. Tooth with a full crown or veneer.
  5. Tooth adjacent to a bridge abutment or crown which, in the opinion of the investigator or dentally qualified designee, could impact study outcomes.
  6. Sensitive tooth with contributing etiologies other than EAR to exposed dentine.
  7. Sensitive tooth not expected to benefit from use of a sensitivity toothpaste, in the opinion of the investigator or dentally qualified designee.
* Participants who, in the opinion of the investigator or designee, are unable to provide appropriate responses to the Labelled Magnitude Scale (LMS) training questions.
* Participants who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Least Square (LS) Mean Change from Baseline in Schiff Sensitivity Score at Day 15 | Baseline (Day 1) and Day 15
  Evaporative (air) sensitivity will be assessed by participant's response to an evaporative (air) stimulus after stimulation of 2 selected test teeth. Response of participant will be scored using Schiff sensitivity scale which ranges from 0-3, where 0=Does not respond to air stimulation; 1=Responds to air stimulus but does not request discontinuation of stimulus; 2=Responds to air stimulus and requests discontinuation or moves from stimulus; 3=Responds to stimulus, considers stimulus to be painful and requests discontinuation of the stimulus. Schiff sensitivity score= average score of the 2 'test teeth' identified at baseline. LS means of change from baseline at Day 15 will be estimated using a Mixed Model with Repeated Measures (MMRM). A decrease in Schiff sensitivity score indicates an improvement.
LS Mean Change from Baseline in Tactile Threshold at Day 15 | Baseline (Day 1) and Day 15
  The tactile sensitivity will be assessed by administrating a constant pressure using a Yeaple probe. At baseline the upper test limit is 20 g and at Day 15, the upper test limit is 80 g. The tactile threshold is the maximum pressure applied without the participant reporting pain or discomfort. The tactile threshold for 2 selected test teeth will be determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gives two consecutives 'yes' responses will be recorded as the tactile threshold. The greater the tactile threshold, the less sensitive the tooth. Tactile threshold= average value for the two 'test teeth' identified at baseline. LS means of change from baseline at Day 15 will be estimated using a MMRM.
Schiff Sensitivity Score at Baseline, Day 2, Day 8, and Day 15 | Baseline (Day 1), Days 2, 8 and 15
  Evaporative (air) sensitivity will be assessed by participant's response to an evaporative (air) stimulus after stimulation of 2 selected test teeth. Response of participant will be scored using Schiff sensitivity scale which ranges from 0-3, where 0=Does not respond to air stimulation; 1=Responds to air stimulus but does not request discontinuation of stimulus; 2=Responds to air stimulus and requests discontinuation or moves from stimulus; 3=Responds to stimulus, considers stimulus to be painful and requests discontinuation of the stimulus. Schiff sensitivity score= average score of the 2 'test teeth' identified at baseline. A decrease in Schiff sensitivity score indicates an improvement.
Tactile Threshold at Baseline, Day 2, Day 8, and Day 15 | Baseline (Day 1), Days 2, 8 and 15
  The tactile sensitivity will be assessed by administrating a constant pressure using a Yeaple probe. At baseline the upper test limit is 20 g and at Day 2, 8 and 15, the upper test limit is 80 g. The tactile threshold is the maximum pressure applied without the participant reporting pain or discomfort. The tactile threshold for 2 selected test teeth will be determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gives two consecutives 'yes' responses will be recorded as the tactile threshold. The greater the tactile threshold, the less sensitive the tooth. Tactile threshold= average value for the two 'test teeth' identified at baseline.
Change From Baseline in Schiff Sensitivity Score at Day 2, Day 8, and Day 15 | Baseline (Day 1), Days 2, 8 and 15
  Evaporative (air) sensitivity will be assessed by participant's response to an evaporative (air) stimulus after stimulation of 2 selected test teeth. Response of participant will be scored using Schiff sensitivity scale which ranges from 0-3, where 0=Does not respond to air stimulation; 1=Responds to air stimulus but does not request discontinuation of stimulus; 2=Responds to air stimulus and requests discontinuation or moves from stimulus; 3=Responds to stimulus, considers stimulus to be painful and requests discontinuation of the stimulus. Schiff sensitivity score= average score of the 2 'test teeth' identified at baseline. Change from baseline will be calculated by subtracting baseline score from the score at the indicated timepoints. A decrease in Schiff sensitivity score indicates an improvement.
Change From Baseline in Tactile Threshold at Day 2, Day 8, and Day 15 | Baseline (Day 1), Days 2, 8 and 15
  The tactile sensitivity will be assessed by administrating a constant pressure using a Yeaple probe. At baseline the upper test limit is 20 g and at Day 15, the upper test limit is 80 g. The tactile threshold is the maximum pressure applied without the participant reporting pain or discomfort. The tactile threshold for 2 selected test teeth will be determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gives two consecutives 'yes' responses will be recorded as the tactile threshold. The greater the tactile threshold, the less sensitive the tooth. Tactile threshold= average value for the two 'test teeth' identified at baseline. Change from baseline will be calculated by subtracting LS mean baseline score from the score at the indicated timepoints.

SECONDARY OUTCOMES:
LS Mean Change from Baseline in Schiff Sensitivity Score at Day 2 and Day 8 | Baseline (Day 1), Days 2 and 8
  Evaporative (air) sensitivity will be assessed by participant's response to an evaporative (air) stimulus after stimulation of 2 selected test teeth. Response of participant will be scored using Schiff sensitivity scale which ranges from 0-3, where 0=Does not respond to air stimulation; 1=Responds to air stimulus but does not request discontinuation of stimulus; 2=Responds to air stimulus and requests discontinuation or moves from stimulus; 3=Responds to stimulus, considers stimulus to be painful and requests discontinuation of the stimulus. Schiff sensitivity score= average score of the 2 'test teeth' identified at baseline. LS means of change from baseline at the indicated timepoints will be estimated using a MMRM. A decrease in Schiff sensitivity score indicates an improvement.
LS Mean Change from Baseline in Tactile Threshold (g) at Day 2 and Day 8 | Baseline (Day 1), Days 2 and 8
  The tactile sensitivity will be assessed by administrating a constant pressure using a Yeaple probe. At baseline the upper test limit is 20 g and at Day 15, the upper test limit is 80 g. The tactile threshold is the maximum pressure applied without the participant reporting pain or discomfort. The tactile threshold for 2 selected test teeth will be determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gives two consecutives 'yes' responses will be recorded as the tactile threshold. The greater the tactile threshold, the less sensitive the tooth. Tactile threshold= average value for the two 'test teeth' identified at baseline. LS means of change from baseline at the indicated timepoints will be estimated using a MMRM.
LS Mean Change from Baseline in Schiff Sensitivity Score at Day 2, Day 8 and Day 15 (Test Versus [Vs] Negative Control) | Baseline (Day 1), Days 2, 8 and 15
  Evaporative (air) sensitivity will be assessed by participant's response to an evaporative (air) stimulus after stimulation of 2 selected test teeth. Response of participant will be scored using Schiff sensitivity scale which ranges from 0-3, where 0=Does not respond to air stimulation; 1=Responds to air stimulus but does not request discontinuation of stimulus; 2=Responds to air stimulus and requests discontinuation or moves from stimulus; 3=Responds to stimulus, considers stimulus to be painful and requests discontinuation of the stimulus. Schiff sensitivity score= average score of the 2 'test teeth' identified at baseline. LS means of change from baseline at the indicated timepoints will be estimated using a MMRM. A decrease in Schiff sensitivity score indicates an improvement.
LS Mean Change from Baseline in Tactile Threshold (g) at Day 2, Day 8 and Day 15 (Test Vs Negative Control) | Baseline (Day 1), Days 2, 8 and 15
  The tactile sensitivity will be assessed by administrating a constant pressure using a Yeaple probe. At baseline the upper test limit is 20 g and at Day 15, the upper test limit is 80 g. The tactile threshold is the maximum pressure applied without the participant reporting pain or discomfort. The tactile threshold for 2 selected test teeth will be determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gives two consecutives 'yes' responses will be recorded as the tactile threshold. The greater the tactile threshold, the less sensitive the tooth. Tactile threshold= average value for the two 'test teeth' identified at baseline. LS means of change from baseline at the indicated timepoints will be estimated using a MMRM.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bristol, Bristol Dental School and Hospital, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.